CLINICAL TRIAL: NCT04195425
Title: Influence of Breastfeeding on Gut Health in Children
Brief Title: Breastfeeding and Gut Health
Acronym: PENSINE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_67; 2019-A01416-51 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2019-12-04; First posted 2019-12-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Gut Health
Keywords: breastfeeding; early nutrition; intestinal microbiota
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cord blood mononuclear cells, meconium/stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of the study is to evaluate the impact of early nutrition on gut health in children. A prospective cohort of newborns will be recruited at birth and followed up to 4 years of age. Information on parent's nutritional habits and life style, breastfeeding duration and child's complementary feeding, will be collected. Cord blood cells and stools will be collected at birth, 6 months, 2 years and 4 years of age for implementing a biological collection. Gut health will be evaluated in children during the first four years of life based on fecal secretory immunoglobulin A (SIgA) and presence of digestive symptoms. Precise data on breastfeeding practices and their short- and medium-term effects on the health of the child, in particular and in an innovative way on gut health, will be obtained.

ELIGIBILITY:
Inclusion Criteria:

For the mother:

* Pregnant woman (>18 years old) followed at the Lille University Jeanne de Flandres Maternity
* Woman who can speak, read and write in French
* Single pregnancy
* Informed consent
* Living in the Lille area

For the father:

* Men >18 years old
* Informed consent

Exclusion Criteria:

For the mother:

* Impossibility to participate to the study follow-up
* Woman under guardianship or curatorship
* Woman involved in another study inconsistent with biological samples collection

For the child after birth:

* Prematurity <37 weeks
* Impossibility to participate to the study follow-up
* Child under judicial protection measure
* Child involved in another study inconsistent with biological samples collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant woman
Study Population: Monocentric cohort including mother/child dyads recruited in a University Maternity
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between exclusive breastfeeding and gut health based on the non-invasive measurement of fecal secretory immunoglobulin A (sIgA) | AT 4 years

SECONDARY OUTCOMES:
Correlation between gut health and the duration of exclusive breastfeeding | A 1 month, 1-2 months, 2-4 months, 4-6 months, 6 months
  defined by the production of Igas in the faeces and the duration of exclusive breastfeeding (1 month, 1-2 months, 2-4 months, 4-6 months, 6 months) collected by mother's interrogation.
Correlation between the mother's feeding habits during pregnancy and the child's gut health during the first 4 years of life | At 6 months, 2 years and 4 years
  Nutritional data collected via the Food Frequency Questionnaire (FFQ) and the mother's obstetric record and Intestinal health of the child during the first 4 years of life evaluated by the production of Igas
Correlation between sIgA and child growth and gastro-intestinal disorders | At 6 months, 2 years and 4 years
  defined by Production of Igas in children and the head circumference, weight and height of the child reported in the health log and the presence of gastrointestinal symptoms evaluated according to the criteria of ROME IV.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Ley, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France

REFERENCES:
- [Derived] Ley D, Beghin L, Morcel J, Flamein F, Garabedian C, Accart B, Drumez E, Labreuche J, Gottrand F, Hermann E. Impact of early life nutrition on gut health in children: a prospective clinical study. BMJ Open. 2021 Sep 6;11(9):e050432. doi: 10.1136/bmjopen-2021-050432. PMID 34489289